CLINICAL TRIAL: NCT06600399
Title: Similarity of Biological Information Captured by (68)Gallium-prostate Specific Membrane Antigen-11 Positron Emission Tomography and Arterial Spin Labeling Perfusion Imaging in Glioblastoma
Brief Title: Correlation Between Prostate-specific Membrane Antigen Positron Emission Tomography and Arterial Spin Labeling Perfusion Imaging in Glioblastoma
Acronym: PSMA，ASL，PET
Status: Completed | Type: Observational
Sponsor: Lanzhou University Second Hospital (Other)
Responsible Party: Principal Investigator, Jing Zhang, chief physician, Lanzhou University Second Hospital
Other Study IDs: JZhang-1990; 23JRRA1625 (Other Grant/Funding Number: the Natural Science Foundation of Gansu Province)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma
Keywords: Prostate-specific membrane antigen; Arterial spin labeling
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — The expression of prostate-specific membrane antigen in glioblastoma multiforme microvascular was analyzed by immunohistochemistry in tissue samples obtained after surgical resection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Correlation between PSMA PET and ASL: The relationship between multimodal images
  Interventions: Diagnostic Test: glioblastoma

INTERVENTIONS:
Diagnostic Test: glioblastoma — All patients underwent conventional MRI, ASL perfusion imaging and 68Ga-PSMA-11 PET/CT examinations within 1 week interval

SUMMARY:
Evaluating the relationship between prostate-specific membrane antigen positron emission tomography and arterial spin labeling perfusion imaging, and the correlation with prostate-specific membrane antigen expressed on glioblastoma microvascular.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or recurrent glioblastoma;
* Adult (≥18 years old);

Exclusion Criteria:

* The patient has a serious underlying disease or mental illness and is unable to cooperate with the imaging examination;
* Have received systematic chemotherapy;
* The image data is of poor or incomplete quality;
* pregnant women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-six patients with newly diagnosed or recurrent glioblastoma who underwent conventional MRI, ASL and PSMA PET were prospectively enrolled
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
The similarity of biological information | 2 week
  Evaluating the similarity of biological information captured by prostate-specific membrane antigen positron emission tomography and arterial spin labeling perfusion imaging in glioblastoma.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: Undecided